CLINICAL TRIAL: NCT02415270
Title: Switching to Reduced Nicotine Content Cigarettes or Reduced Reactive Oxygen/Reactive Nitrogen Species Cigarettes in Smokers
Brief Title: Switching to Reduced Oxidant or Nicotine Content Cigarettes in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John P. Richie, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001996; 5P50DA036107-02 (NIH)
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Tobacco Smoking Behavior
MeSH Terms: conditions — Smoking | interventions — Menthol; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Reduced Nicotine Cigarettes (Experimental): Participants will be randomized to receive low nicotine cigarettes to replace their usual high nicotine brand.
  Interventions: Other: Reduced Nicotine Cigarettes
- Reduced ROS/RNS (Experimental): Participants will be randomized to receive Reduced Oxidative/Nitrogen Species (ROS/RNS) cigarettes to replace their usual cigarettes.
  Interventions: Other: Reduced ROS/RNS
- Control Group (Placebo Comparator): Participants will be assigned to continue smoking their usual brand of cigarettes.
  Interventions: Other: Control

INTERVENTIONS:
Other: Reduced Nicotine Cigarettes — Human topography data will show if smokers smoke their cigarettes differently from baseline following randomization. Select biosamples of participants will be used to analyze how biomarkers differ among groups
  Other Names: Cigarette contains .28mg (.29mg/menthol) of nicotine
  Arms: Reduced Nicotine Cigarettes
Other: Reduced ROS/RNS — Human topography data will show if smokers smoke their cigarettes differently from baseline following randomization. Select biosamples of participants will be used to analyze how biomarkers differ among groups
  Other Names: Cigarette to be determined by lab experiment
  Arms: Reduced ROS/RNS
Other: Control — Human topography data will show if smokers change the way they smoke due to being in a research study. Select biosamples of participants will be used to analyze how biomarkers differ among groups
  Arms: Control Group

SUMMARY:
The overall objectives of this clinical study are to determine in smokers the short term effects of switching to tobacco products that deliver low levels of nicotine or reactive oxygen/nitrogen species (ROS/RNS) on smoking behavior and biomarkers of tobacco smoke exposure and oxidative stress.

DETAILED DESCRIPTION:
Researchers at Penn State Hershey are seeking healthy adult cigarette smokers between 21-65 who smoke any of the following brands on a regular basis: Marlboro Red, Marlboro Menthol, Pall Mall Red, Pall Mall Menthol, Kool Menthol, Salem Menthol, L&M Menthol, Pyramid Red, Newport Red, Newport Menthol.

If you smoke one of these brand styles on a regular basis you may be eligible to participate in a compensated short term study on health and smoking behavior at Penn State Hershey Medical Center.

Study participation lasts 22 days, with 4 study visits at the Medical Center. Smokers are asked to use their usual brand for one week and then switch to 1 of 3 brands for the remaining two weeks. The three brands participants are randomly assigned to after the first week of participation are either Group 1. reduced nicotine content cigarette (Spectrum Research Cigarettes) or Group 2. reduced oxidant cigarette (American Spirit) or assigned to Group 3. usual brand. Whichever group you are assigned to, you will be asked to smoke only these until the end of the study. All cigarettes following visit 1 will be provided free of charge.

Study overview:

Visit 1/ Duration: 60 minutes Provide a blood and urine sample Complete a 20 minute interview Use a simple, hand held smoking device to smoke all cigarettes for 2 days Collect cigarette butts on 1 day

Visit 2: Randomized Phase /Duration: 20-30 minutes Provide a blood and urine sample Complete a 10 minute interview Use a simple, hand held smoking device to smoke all cigarettes for 2 days Collect cigarette butts on 1 day

Visit 3/ Duration: 20-30 minutes Provide a blood and urine sample Complete a 10 minute interview Use a simple, hand held smoking device to smoke all cigarettes for 2 days Collect cigarette butts on 1 day

Visit 4/ Duration: 20-30 minutes Provide a blood and urine sample Complete a 10 minute interview Sign compensation form

For information on additional tobacco studies being conducted at Penn State Hershey, please call 1-844-207-6392

*This research is being conducted under the investigator John Richie at Penn State Hershey; 500 University Drive Hershey, PA

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Smoke 10 cigarettes/day or more for at least one year
* Read and write in English
* Menthol and nonmenthol smokers who use relatively high nicotine and ROS/RNS cigarettes
* Able to understand and provide consent to study procedures
* Plan to live in the local area for the next month
* Women not pregnant or nursing and taking steps to avoid pregnancy
* No quit attempt in the last one months and not planning to quit in the next month

Exclusion Criteria:

* Currently pregnant or nursing
* Unstable or significant medical condition, such as COPD or kidney failure, that is likely to affect biomarker data
* Use of non-cigarette nicotine delivery product in the past week (included cigars, pipes, chew, snus, hookah, e-cig, and marijuana)
* Currently reducing or planning to reduce cigarette consumption in the next month
* Use of smoking cessation medicine in the past 3 months
* History of difficulties providing blood samples: fainting, poor veins, anxiety, etc.
* Uncontrolled serious psychotic illness or substance abuse or inpatient treatment for these in the last 6 months (substance abuse includes weekly, almost daily or daily use of other illegal drugs and prescription drugs that are not being used for medically prescribed purposes or alcohol abuse that would hinder the participant's ability to participate)
* Significant medical condition, i.e. stroke, MI, cancer, in the last month
* Currently using illegal drugs

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Smoking Topography | 8 days
  measures of smoking topography include parameters such as puff volume, frequency and intensity as measured using a smoking topography instrument.

SECONDARY OUTCOMES:
Biomarkers of oxidative stress | 4 times over the 22 day study period
  biomarkers of oxidative stress are as followed: glutathionylated and cysteinylated proteins in blood and F2-isoprostanes and 8-hydroxydeoxyguanosine (8-OHdG).

CONTACTS AND LOCATIONS:
Overall Officials: John Richie, Ph.D, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time we have no plan for sharing, however if need should arise, then sharing may be a possibility.